CLINICAL TRIAL: NCT06863662
Title: Efficacy and Safety of the Fixed-Dose Combination of Etoricoxib / Tizanidine Versus Etoricoxib in the Treatment of Patients With Acute Low Back Pain Associated to Muscle Spasm
Brief Title: Efficacy and Safety of Etoricoxib/Tizanidine Versus Etoricoxib for Acute Low Back Pain Associated to Muscle Spasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30951-III-23(1)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Acute Low-back Pain; Muscle Spasm; Back Pain
Keywords: Acute Low-back Pain; Back pain with muscle spams; Etoricoxib; Tizanidine
MeSH Terms: conditions — Spasm; Back Pain | interventions — Etoricoxib; tizanidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib+Tizanidine (Experimental): Administered orally, 1 sachet a day for 7 days.
  Interventions: Drug: Etoricoxib + Tizanidine fixed dose
- Etoricoxib (Active Comparator): Administered orally, 1 sachet a day for 7 days.
  Interventions: Drug: Etoricoxib fixed dose

INTERVENTIONS:
Drug: Etoricoxib + Tizanidine fixed dose — One sachet with 120 mg / 4 mg, dissolved in 100 mL of water
  Other Names: Etori + Tiza
  Arms: Etoricoxib+Tizanidine
Drug: Etoricoxib fixed dose — One sachet with 120 mg, dissolved in 100 mL of water
  Other Names: Etori
  Arms: Etoricoxib

SUMMARY:
This is a Phase III, longitudinal, multicenter, randomized, double-blind clinical trial. The aim of the study is to evaluate the efficacy and safety of a fixed-dose combination of etoricoxib and tizanidine compared to etoricoxib alone in patients with acute low back pain associated with muscle spasms.

DETAILED DESCRIPTION:
Researchers will compare the efficacy of a fixed-dose combination of etoricoxib and tizanidine versus etoricoxib alone in the treatment of acute low back pain associated with muscle spasms. Efficacy will be assessed by evaluating the average change in pain among patients who report improvement over the 7-day follow-up period. Adverse events related to the interventions will be recorded throughout the study.

Participants will:

* Be randomized into one of two intervention groups (Group A or Group B).
* Attend three in-person clinic visits: Day 0 (baseline), Day 3, and Day 7 of follow-up.
* Receive follow-up phone calls on Days 1 and 5.
* Be allowed to take 500 mg of acetaminophen as rescue medication if needed, with prior authorization from the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Diagnosis of acute low back pain, either as a first-time episode or following a previous episode within the past 6 months, with a duration not exceeding 6 weeks.
* Pain associated with lumbar muscle spasm, assessed through physical examination (muscle hypertonia and/or reflex scoliosis) and clinical history.
* Patient reports moderate to severe pain intensity (VAS ≥ 40 mm).
* Patients with a Neuropathic Pain Questionnaire (DN4) score < 4.
* For women of childbearing age who are sexually active, the use of an acceptable contraceptive method (barrier and/or hormonal) as determined by the investigator.
* At the discretion of the Principal Investigator (PI) or treating physician, the patient is eligible for treatment with the investigational product and may benefit from it.

Exclusion Criteria:

* Patients with a history of hypersensitivity to any components of the investigational product (Etoricoxib/Tizanidine) or their derivatives (as reported in the medical history and clinical interview).
* Patients participating in another clinical trial involving an investigational treatment or who have participated in one within the past 2 weeks before the study begins.
* Patients whose participation in the study may be influenced (e.g., employment relationship with the research center or sponsor, vulnerable populations, etc.).
* Patients for whom the investigational drug is contraindicated for medical reasons.
* Positive pregnancy test, pregnant women, breastfeeding women, or those planning a pregnancy during the study period.
* Significant history of gastrointestinal disorders (e.g., active gastric ulcer, Crohn's disease, ulcerative colitis, etc.).
* Prior treatment with opioids and/or NSAIDs, including COX-2 inhibitors, as reported in the medical history within 48 hours before study enrollment.
* Patients with a history of congestive heart failure: NYHA class II-IV.
* Concomitant use of potent CYP1A2 inhibitors (e.g., fluvoxamine, ciprofloxacin, etc.).
* History of alcohol or drug abuse within the past year.
* Patients with a history of established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease (including patients who have recently undergone coronary revascularization procedures or angioplasty).
* Patients with a history of seizure disorders, status epilepticus, or grand mal seizures.
* History of liver disease classified as Child-Pugh A, B, or C, as reported in the medical history or clinical interview.
* History of acute or severe renal failure (glomerular filtration rate <30 ml/min/1.73 m²), as reported in the medical history or clinical interview.
* Patients with a history of chronic musculoskeletal pain (e.g., fibromyalgia, Paget's disease, cancer-induced metastatic bone pain).
* Patients diagnosed with low back pain due to a history of major trauma within the past 12 months (e.g., vertebral fracture, post-traumatic spondylolisthesis), a visceral disorder (e.g., dysmenorrhea, history of endometriosis), or a neuropathic component.
* At the physician's discretion, any disease that affects prognosis and prevents outpatient management, which must be evaluated by the principal investigator to determine the subject's eligibility.
* History or presence of any disease or condition that, in the investigator's opinion, could pose a risk to the patient or confound the efficacy and safety assessment of the investigational product.
* Patients with symptoms suggesting an active COVID-19 infection (e.g., fever, cough, dyspnea) and/or contact with a suspected or confirmed COVID-19 case in the last 14 days.
* Oncology patients (except for basal cell skin cancer) or those with severe illnesses who, in the investigator's opinion, have a severe prognosis or a life expectancy of less than one year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage change in pain intensity, as measured by the Visual Analog Scale (VAS), on Days 1, 3, 5, and 7 of follow-up relative to baseline, within each treatment group. | 7 days
  The Visual Analog Scale (VAS) for pain is a straight line anchored by two descriptors: one end indicating no pain and the other representing the worst pain imaginable. The investigator will administer the VAS at each study visit to assess pain intensity. At the end of the clinical trial, the percentage change in pain scores from baseline will be calculated and compared between treatment groups.
Number of participants reporting treatment-related adverse events, as documented in the patient diary. | 7 days
  To describe the frequency, intensity, and causality of adverse events reported during the clinical trial, stratified by treatment group. Adverse events will be recorded by patients in their diary logs. Each event will be monitored and followed up at the discretion of the investigator.

SECONDARY OUTCOMES:
Analyze the percentage change in pain intensity, as measured by the Visual Analog Scale (VAS), on Days 1, 3, 5, and 7, compared to baseline, within and between each treatment group. | 7 days
  The Visual Analog Scale (VAS) for pain is a straight line anchored by two descriptors: one end represents the absence of pain, and the other indicates the worst pain imaginable. The investigator will administer the VAS at each study visit to assess pain intensity. At the end of the clinical trial, the percentage change in pain scores from baseline will be calculated and compared across treatment groups. Patients will attend in-person visits on Days 0, 3, and 7 of follow-up, and the investigator will conduct follow-up phone calls on Days 1 and 5.
Compare the proportion of patients in each treatment group who achieve a ≥30% reduction in pain intensity, as measured by the Visual Analog Scale (VAS), on Days 1, 3, 5, and 7 relative to baseline. | 7 days
  The Visual Analog Scale (VAS) for pain is a unidimensional tool consisting of a straight line anchored by two descriptors: one end indicating "no pain" and the other representing "the worst pain imaginable." The investigator will administer the VAS at each study visit to assess pain intensity. The proportion of patients achieving a reduction in pain of more than 30% from baseline will be recorded and compared across treatment groups on Days 1, 3, 5, and 7.
Compare the proportion of patients in each treatment group who achieve a ≥50% reduction in pain intensity, as measured by the Visual Analog Scale (VAS), on Days 1, 3, 5, and 7 relative to baseline. | 7 days
  The Visual Analog Scale (VAS) for pain is a straight line anchored by two descriptors: one end represents the absence of pain, and the other indicates the worst pain imaginable. The investigator will administer the VAS at each study visit to evaluate pain intensity. The proportion of patients achieving a pain reduction greater than 30% from baseline will be documented and compared across treatment groups on Days 1, 3, 5, and 7.
Determine the follow-up time point at which each treatment group demonstrates the greatest reduction in pain intensity, as measured by the Visual Analog Scale (VAS). | 7 days
  The Visual Analog Scale (VAS) for pain is a unidimensional measurement tool represented by a straight line anchored by two descriptors: one end indicating "no pain" and the other representing "the worst pain imaginable." The investigator will administer the VAS at each study visit to assess the patient's pain intensity.
Compare the proportion of patients in each treatment group according to the severity of lumbar muscle spasm, as assessed by the Investigator's Global Subjective Assessment. | 7 days
  The investigator will assess the severity of lumbar muscle spasm using a global subjective scale, which will also allow evaluation of the muscle's response to movement following administration of the study treatment.
Assess and compare the degree of physical disability caused by acute low back pain, as measured by the Oswestry Disability Questionnaire, on Days 3 and 7 in each treatment group, relative to baseline. | 7 days
  The Oswestry Disability Questionnaire is designed to assess how back pain affects a patient's ability to perform daily activities. It categorizes quality of life into five levels: no disability, mild disability, moderate disability, severe disability, and complete disability. The degree of disability will be assessed and compared between treatment groups.
Assess and compare the degree of disability in performing daily activities due to low back pain, as reported using the Roland-Morris Disability Questionnaire, on Days 3 and 7 in each treatment group, relative to baseline. | 7 days
  The Roland-Morris Disability Questionnaire is designed to assess functional mobility and limitations in daily activities due to low back pain. It consists of 24 items, with higher scores indicating a greater degree of disability. A maximum score of 24 reflects the most severe disability. The degree of disability will be assessed and compared between treatment groups.

OTHER OUTCOMES:
Report the percentage of therapeutic adherence on Day 7 of the intervention, in each treatment group. | 7 days
  Therapeutic adherence will be defined by the principal investigator. Adherence will be considered adequate when the patient has taken ≥80% of the prescribed doses by the time of the corresponding evaluation.
Report the number of patients in each treatment group who require the use of rescue medication during the clinical trial. | 7 days
  The designated rescue medication will be acetaminophen 500 mg. If a patient feels the need for rescue medication, they must contact the study physician. The physician will assess the patient's pain using the Visual Analog Scale (VAS) via telephone. If deemed appropriate, the physician will authorize the use of the rescue medication.
Report the number of patients who experience therapeutic failure during the study, stratified by treatment group. | 7 days
  Therapeutic failure will be defined by the principal investigator following a medical consultation. The following criteria must be met: a decrease of less than 10 mm or an increase in pain intensity on the Visual Analog Scale (VAS) compared to baseline, along with a treatment adherence rate of ≥80%.

CONTACTS AND LOCATIONS:
Overall Officials: Lilia E Acevedo-Rojas, MD, Principal Investigator — Oaxaca Site Management Organization, S.C.; Mauricio Flores-Araujo, MD, Principal Investigator — Mérida/ Investigación Clínica; Salvador Perez-Jaime, MD, Principal Investigator — Centro de Investigación Médica Aguascalientes (CIMA)
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgartner PC, Haynes RB, Hersberger KE, Arnet I. A Systematic Review of Medication Adherence Thresholds Dependent of Clinical Outcomes. Front Pharmacol. 2018 Nov 20;9:1290. doi: 10.3389/fphar.2018.01290. eCollection 2018. PMID 30524276
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Kovacs FM, Llobera J, Gil Del Real MT, Abraira V, Gestoso M, Fernandez C, Primaria Group KA. Validation of the spanish version of the Roland-Morris questionnaire. Spine (Phila Pa 1976). 2002 Mar 1;27(5):538-42. doi: 10.1097/00007632-200203010-00016. PMID 11880841
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Perez C, Galvez R, Huelbes S, Insausti J, Bouhassira D, Diaz S, Rejas J. Validity and reliability of the Spanish version of the DN4 (Douleur Neuropathique 4 questions) questionnaire for differential diagnosis of pain syndromes associated to a neuropathic or somatic component. Health Qual Life Outcomes. 2007 Dec 4;5:66. doi: 10.1186/1477-7525-5-66. PMID 18053212
- [Background] van Tulder MW, Touray T, Furlan AD, Solway S, Bouter LM; Cochrane Back Review Group. Muscle relaxants for nonspecific low back pain: a systematic review within the framework of the cochrane collaboration. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1978-92. doi: 10.1097/01.BRS.0000090503.38830.AD. PMID 12973146
- [Background] Pallay RM, Seger W, Adler JL, Ettlinger RE, Quaidoo EA, Lipetz R, O'Brien K, Mucciola L, Skalky CS, Petruschke RA, Bohidar NR, Geba GP. Etoricoxib reduced pain and disability and improved quality of life in patients with chronic low back pain: a 3 month, randomized, controlled trial. Scand J Rheumatol. 2004;33(4):257-66. doi: 10.1080/03009740410005728. PMID 15370723